CLINICAL TRIAL: NCT07130253
Title: Efficacy of Vonoprazan-based Rescue Therapy for H. Pylori Eradication
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202506082MINA
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: HELICOBACTER PYLORI INFECTIONS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empirical vonoprazan-based therapy (Experimental)
  Interventions: Drug: Vonoprazan based ET
- Susceptibility-guided vonoprazan-based therapy (Active Comparator)
  Interventions: Drug: Vonoprazan based SGT

INTERVENTIONS:
Drug: Vonoprazan based ET — Empirical therapy Based on drug history: Levofloxacin sequential therapy or bismuth quadruple therapy (10 or 14 days) or quadruple therapy
  Arms: Empirical vonoprazan-based therapy
Drug: Vonoprazan based SGT — Susceptibility testing guided therapy Based onsusceptibility test:Levofloxacin sequential therapy or bismuth quadruple therapy (10 or 14 days) or rifabutin quadruple therapy
  Arms: Susceptibility-guided vonoprazan-based therapy

SUMMARY:
1. This study aims to compare the efficacy of empirical vonoprazan-based therapy versus susceptibility-guided vonoprazan-based therapy for third-line eradication of H. pylori.
2. We also plan to explore the impact of eradication therapy on gut microbiota, fecal antibiotic resistance, and metabolic parameters before and after treatment.

DETAILED DESCRIPTION:
Methods:

* Study design: Open-labeled, randomized controlled trial
* Participants: A total of 220 patients who have failed at least two previous H. pylori eradication treatments will be enrolled.

Determination of antibiotic resistance of H. pylori: Agar dilution test will be used to determine the minimum inhibitory concentrations of levofloxacin, tetracycline, rifabutin, and clarithromycin to guide the selection of antibiotics.

Treatment regimens and assignment: Eligible patients will be randomized to receive either one of the treatments (A) Empirical vonoprazan-based therapy or (B) Susceptibility-guided vonoprazan-based therapy

Outcome Measurement:

Primary End Point: Eradication rate by intention-to-treat analysis. Secondary End Point: 1. Eradication rate by per-protocol analysis; 2. Frequency of adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. Helicobacter pylori infected individuals who have failed at least two previous eradication therapies.
2. Willing to undergo third-line eradication therapy.
3. Subjects must be 20 years of age or older.

Exclusion Criteria:

1. History of gastrectomy.
2. Individuals unsuitable for the study medication, such as those with a history of allergy or severe adverse reactions to the study drugs, quinolone or fluoroquinolone antibiotics, or women who are pregnant or breastfeeding.
3. Presence of severe acute or chronic diseases such as renal failure, liver cirrhosis, incurable malignant tumors, or a history of aortic aneurysm or dissection.
4. Patients with chronic hepatitis (AST or ALT > 100 U/L).
5. Unwillingness to comply with the treatment plan or sign the informed consent form.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Eradication rate by intention-to-treat analysis | 6-8 weeks
  Eradication rate will be determined by urea breath test at least 6 weeks aftercompletion of treatment.

SECONDARY OUTCOMES:
Eradication rate by per-protocol analysis and Frequency of adverse effects. | 6-8 weeks
  Eradication rate will be determined by urea breath test at least 6 weeks aftercompletion of treatment. A standard interview and questionaire will be used to assess the adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Ming Liou, MD, PhD, Study Director — National Taiwan University Hospital; Mei-Jyh Chen, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No